CLINICAL TRIAL: NCT00657098
Title: Mabtornib Protocol.Vascular, Metabolic and Hormonal Effects of Angiogenesis Inhibitors and Epidermal Growth Factor Receptor Inhibitors
Brief Title: Side Effects of Vascular Endothelial Growth Factor (VEGF) and Epidermal Growth Factor Receptor (EGFR) Directed Therapy
Acronym: Mabtornib
Status: Terminated | Type: Observational
Why Stopped: slow inclusion rate
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 2007/203
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Malignancies
Keywords: Side effects; Angiogenesis inhibitors; Epidermal growth factor receptor inhibitors; Tyrosinekinase inhibitors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma Urine DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation

SUMMARY:
Angiogenesis inhibitors and EGFR inhibitors not only have anti tumor activity but also modify physiological processes. This study evaluates effects on vascular function, endocrine function and metabolism. Changes in these parameters will be analysed for predictive value for treatment efficacy.

DETAILED DESCRIPTION:
Background

In recent years, multiple new agents have been developed that inhibit angiogenesis and the epidermal growth factor receptor (EGFR) signalling pathway.

The cell signalling routes that are inhibited by these agents however are not only active in tumour formation but are also involved in physiological processes in normal tissue and organs. This means that these drugs do not only have an anti tumour effect but also modify several physiological processes that lead to side effects. Little is known about these side effects that generally are less severe than side effects of cytotoxic chemotherapy, but because targeted therapy is often administered for prolonged periods of time, these side effects can seriously affect quality of life.

Objectives

Primary objectives

1. To determine the characteristics, frequency and severity of vascular, metabolic and hormonal side effects of angiogenesis and EGFR inhibitors.

Secondary objectives

1. To investigate if steroid profile, indol profile, concentrations of catecholamines and metanephrines or thyroid antibodies change during treatment with angiogenesis and EGFR inhibitors.
2. To investigate if known biomarkers change during treatment.
3. To investigate whether vascular function changes during treatment with angiogenesis and EGFR inhibitors.
4. To determine if changes in skin autofluorescence and development of AGE's occur during treatment with angiogenesis and EGFR inhibitors.
5. To determine whether changes in factors mentioned under secondary objectives 1-4 are correlated with side effects of targeted therapy and/or response to angiogenesis and EGFR inhibitors.
6. To evaluate if polymorphisms in genes involved in pathways mentioned under 1-4 associate with toxicity and efficacy of angiogenesis and EGFR inhibitors.

Study design and population

This is a prospective, explorative observational cohort study in patients treated with angiogenesis or EGFR inhibitors. Concomitant chemotherapy, immunotherapy or radiotherapy is allowed. Patients must be 18 years or older at start of treatment and must be willing to give written informed consent.

Primary study parameters

Patients will be evaluated for vascular changes by measuring

* 24-hour ambulatory blood pressure
* nail fold capillary microscopy
* skin autofluorescence at 3 time points: before start of treatment, and after 3 and after 6 weeks of treatment. Patients will also be asked to measure their blood pressure at home twice a day, for 6 weeks. Metabolic and hormonal changes and investigation of biomarkers will be done by blood and urine analyses every 3 weeks for the first 3 months, every 6 weeks up to 6 months and every 3 months thereafter.

Changes in vascular, hormonal and metabolic status will be related to clinical side effects and to response to treatment.

Secondary study parameters

When clinically relevant differences in side effects and response to treatment are found among patients treated with the same agent, DNA analysis will be carried out to investigate if changes in candidate genes are related to these differences.

Burden and risks associated with participation, benefit and group relatedness

The minimal invasive tests will be performed during routine outpatient visits. As far as known no serious adverse events are linked to the described study procedures. With this study we hope to get insight into the characteristics, frequency, severity and underlying mechanisms of angiogenesis and EGFR inhibitor induced vascular, metabolic and hormonal side effects and to find usable surrogate markers for efficacy of treatment. Eventually, this may contribute to the early detection of vascular, metabolic and hormonal changes, to the design of intervention strategies for side effects and to better patient selection for angiogenesis and EGFR inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will start with an angiogenesis inhibitor or EGFR inhibitor
* Concomittant chemotherapy, immunotherapy or radiotherapy is allowed
* Age above 18 years at start of treatment
* Willingness to give written informed consent

Exclusion Criteria:

* Unable to give written informed consent
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be treated with angiogenesis inhibitors or EGFR inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2008-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Characteristics, frequency and severity of vascular, metabolic and hormonal side effects of angiogenesis and EGFR inhibitors. | after 3 and after 6 weeks of treatment
  Vascular function tests at baseline, after 3 and after 6 weeks of treatment, blood and urine measurements as long as treatment is continued.

SECONDARY OUTCOMES:
DNA analysis | day -7 till day -1

CONTACTS AND LOCATIONS:
Overall Officials: Jourik A Gietema, MD/PhD, Principal Investigator — University Medical Center Groningen, The Netherlands
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands